CLINICAL TRIAL: NCT07255014
Title: Impact of Epidural on Trauma of the Genital Tract During Peripartum
Status: Completed | Type: Observational
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head Physician of Clinical Trial Unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-PeriTRAU
Record Dates: First submitted 2025-06-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Peripartum Genital Tract Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deliveries with epidural analgesia
  Interventions: Other: Data collection from medical files
- Deliveries without epidural analgesia
  Interventions: Other: Data collection from medical files

INTERVENTIONS:
Other: Data collection from medical files — Data collection from medical files

SUMMARY:
Peripartum genital tract injuries (PVT) are common after vaginal delivery and can lead to physical, psychological, and functional sequelae. While several risk factors have been established in the literature, the link between epidural analgesia and these injuries remains controversial. The primary objective of this study was to evaluate the impact of epidural analgesia on the occurrence of PVT. Secondary objectives were to examine its association with instrumentation, episiotomy, and induction of labor, to identify independent risk factors for PVT, and to develop a predictive model for the risk of these injuries.

ELIGIBILITY:
Inclusion Criteria:

Vaginal delivery within the CHU Brugmann Hospital, from January 1 2020 till December 31 2002

Exclusion Criteria:

* Incomplete medical files
* Delivery before 25 weeks of pregnancy
* Out of Hospital delivery
* Medical termination of pregnancy (MTP)
* Cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women giving birth by vaginal delivery within the CHU Brugmann Hospital, from January 1 2020 till December 31 2002
Sampling Method: Non-Probability Sample
Enrollment: 8516 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Rate of peripartum genital tract trauma | At delivery
  Peripartum genital tract trauma is defined as any obstetric injury occurring during vaginal delivery, including perineal tears, episiotomies, and uterine ruptures.
Type of peripartum genital tract trauma | At delivery
  Distribution and severity of trauma (perineal tears from D1 to D4 according to OMS CIM-10 classification, D1 being superficial damage, versus episiotomies versus uterine ruptures).

SECONDARY OUTCOMES:
Instrumentation rate | At delivery
  Use of forceps, suction cup, spatulas.
Labor induction rate | At delivery
  Labor induction

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Javad BIDGOLI, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium